CLINICAL TRIAL: NCT02472288
Title: Multicenter, Randomised Controlled Trial of Electroacupuncture Versus Sham Electroacupuncture for Urinary Retention of Poststroke Patients: a Study Protocol
Brief Title: Electroacupuncture on Post-stroke Urinary Retention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolling participants
Sponsor: Kyunghee University (Other)
Collaborators: Daejeon University (Other); DongGuk University (Other)
Responsible Party: Principal Investigator, Lee Eui-ju, Professor, Kyunghee University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015008
Record Dates: First submitted 2015-06-09; First posted 2015-06-15 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Urinary Retention; Stroke, Complication
Keywords: urinary retention; poststroke; electroacupuncture; randomized controlled trial; effectiveness; safety
MeSH Terms: conditions — Urinary Retention; Stroke | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electroacupuncture (EA) group (Experimental): 1. Electroacupuncture therapy (10 sessions in total, 5 per a week, 2 weeks)
  2. BL31, BL32, BL33, and BL34 (total 8 acupoints, bilateral)
  3. 20 minutes duration, middle frequency (30 Hz) of electrical stimulation
  4. conventional treatments permitted
  Interventions: Device: Electroacupuncture (EA)
- Sham group (Sham Comparator): 1. Non-penetrating Park sham electroacupuncture treatment (10 sessions in total, 5 per a week, 2 weeks)
  2. BL31, BL32, BL33, and BL34 (total 8 acupoints on the right and left sides)
  3. 20 minutes duration, undelivered electrostimulation of middle frequency (30 Hz)
  4. conventional treatments permitted
  Interventions: Device: Sham electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture (EA) — The EA group receives 10 sessions of EA therapy (5 per a week, 2 weeks). After inserting needles by 5-10 mm (stainless steel, 0.25 mm in diameter and 4.0 mm in length, Dong Bang Acupuncture Inc., Korea) using the Park sham guide tube on the 8 points (BL31, BL32, BL33, and BL34, bilateral sides), de qi response is elicited. The electrical stimulation is then presented for 20 minutes by middle frequency (30 Hz) (STN-111, Stratek, Korea). Conventional treatments (western/traditional herbal medications, rehabilitation, or acupuncture without electro-stimulation for stroke, and western/traditional herbal medications or acupuncture without electro-stimulation for urinary retention) are allowed during the intervention period. The practitioner should have over 1-year clinical experiences.
  Arms: Electroacupuncture (EA) group
Device: Sham electroacupuncture — The patients in sham group receive totally 10 sessions of the sham EA (5 sessions per a week, for 2 weeks). Non-penetrating needles of Park sham device are implemented on the bilateral points of BL31, BL32, BL33, and BL34 (total 8 acupoints). Then, the electro-stimulation is presented for 20 minutes by middle frequency (30 Hz) (STN-111, Stratek, Korea), even though the electrical stimulation is not delivered through the skin. Conventional treatments for stroke and urinary retention along with EAT are not eliminated. It is also necessary for the practitioner with more than 1-year experiences on the clinical field.
  Arms: Sham group

SUMMARY:
This study aimed to evaluate the effectiveness of adjuvant electroacupuncture therapy for the post-stroke patients with urinary retention under conventional treatments, compared with sham electroacupuncture.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged over 19
* Patients diagnosed with stroke (cerebral hemorrhage or infarction) based on the CT or MRI examination
* Those whose onset is within 2 years
* Those who have urinary retention after stroke onset (every PVR result is equal or more than 100ml on the 2 consecutive tests)
* Those who signed on the informed consent form

Exclusion Criteria:

* Patients who have any bleeding disorders based on medical history hearing
* Patients who have ever had any medical procedures or surgeries for peripheral vascular diseases based on medical history hearing
* Patients who have any psychiatry disorders based on medical history hearing
* Patients who have any severe diseases in lower urinary tract symptom based on medical history hearing
* Patients who have any acute or chronic infectious diseases in lower urinary tract symptom based on medical history hearing
* Acute stage stroke patients (onset within 1 week) whose Glasgow Coma Scale ≤ 8
* Patients who have fear about acupuncture
* Patients who have changed medications for urinary retention or relevant symptoms, such as urinary incontinence drugs or diuretics, within 3 days
* Female who diagnosed with pregnancy by urinalysis
* Those who primary or sub investigators judge not to be suitable for the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change of daily PVR (Postvoid Residual) urine ratios between the baseline and the endpoint | Day 0 (baseline), Day 14(endpoint)
  * daily PVR ratio = daily PVR urine volume / (daily PVR urine volume + self voiding volume)
  * Baseline measurement: daily PVR ratio for 24 hours on the day before the first intervention day Endpoint measurement: daily PVR ratio for 24 hours within 3 days after the last intervention day
  * If more than 7 sessions of EA or sham EA are completed and urinary tract is not infected at the end, then the urine volume is measured on the next day of the last intervention.
  * If more than 7 sessions of EA or sham EA are completed and urinary tract is infected at the end, then the urine volume is measured on the 3rd day of the last intervention after anti-infection treatment is carried out for 48 hours.

SECONDARY OUTCOMES:
Urinary tract infection (UTI) | Day 14(endpoint)
  After 7-10 sessions of the EA or sham EA, patients get urinalysis to figure out whether UTI exists. If a patient has UTI, he/she gets antibiotics for 48 hours. When no UTI is found with reexamination of urinalysis, then daily PVR is going to be assessed and included in the final ITT (Intention To Treat) analysis. Otherwise, the data from the patients will be included only in the PP (Per Protocol) analysis.
Korean version of Qualiveen Questionnaire (K-QQ) | Day 0 (baseline), Day 14(endpoint)
  * The disease-specific QoL (quality of life) assessment scale for neurogenic bladder
  * Consisting of 30 items and each item is scored by 0 to 4. (The higher score in K-QQ is, the lower QoL of the patients is.)
  * The reliability and validity of K-QQ has been acquired in the previous studies.
  * If more than 7 sessions of EA or sham EA are completed and urinary tract is not infected at the end, then K-QQ is measured on the next day of the last intervention.
  * If more than 7 sessions of EA or sham EA are completed and urinary tract is infected at the end, then K-QQ is measured on the 3rd day of the last intervention after anti-infection treatment is carried out for 48 hours.
Korean version of International Prostate Symptom Scale (K-IPSS) | Day 0 (baseline), Day 14(endpoint)
  * Assessment tool for symptoms in lower urinary tract
  * Consisting of 7 items (0 to 5 scores)
  * If more than 7 sessions of EA or sham EA are completed and urinary tract is not infected at the end, then K-IPSS is measured on the next day of the last intervention.
  * If more than 7 sessions of EA or sham EA treatment are completed and urinary tract is infected at the end, then K-IPSS is measured on the 3rd day of the last intervention after anti-infection treatment is carried out for 48 hours.
Blinding Index (BI) | Day 14(endpoint)
  * Assessment of patients' blinding
  * Patients are asked which group you think you belong to during the study, and they selects one of the options, EA group, sham group, or Not knowing.
Frequencies of urination and urinary incontinence | Day 0 (baseline), Day 14(endpoint)
  * Record of the frequencies of urination and urinary incontinence by urinary diary
  * 1 day before the first intervention and another day after the last intervention
  * Mean change between post- and pre-treatments in EA group comparing with the sham group
Adverse events | Every treatment visit (5 times during Day 1~Day 7 & 5 times during Day 8~Day 14)
  * Ask any adverse events after EA or sham interventions and record them in case report forms
  * Evaluate the severity, seriousness, and relevance to the study

OTHER OUTCOMES:
Diabetes mellitus (DM) and benign prostatic hyperplasia (BPH) | Day 0 (baseline)
  Check of diabetes mellitus (DM) and benign prostatic hyperplasia (BPH) in medical history.

CONTACTS AND LOCATIONS:
Overall Officials: Euiju Lee, Ph.D., Principal Investigator — Kyunghee University
Locations (3):
- South Korea (3):
  - Cheonan Korean Medicine Hospital of the Daejeon University, Cheonan, Chungcheongnam-do
  - Dongguk University Ilsan Oriental Hospital, Goyang-si, Gyeonggi-do
  - Kyung Hee University Korean Medicine Hospital, Seoul

REFERENCES:
- [Background] Kong KH, Young S. Incidence and outcome of poststroke urinary retention: a prospective study. Arch Phys Med Rehabil. 2000 Nov;81(11):1464-7. doi: 10.1053/apmr.2000.9630. PMID 11083349
- [Background] Wu J, Baguley IJ. Urinary retention in a general rehabilitation unit: prevalence, clinical outcome, and the role of screening. Arch Phys Med Rehabil. 2005 Sep;86(9):1772-7. doi: 10.1016/j.apmr.2005.01.012. PMID 16181941
- [Background] Wu P, Mills E, Moher D, Seely D. Acupuncture in poststroke rehabilitation: a systematic review and meta-analysis of randomized trials. Stroke. 2010 Apr;41(4):e171-9. doi: 10.1161/STROKEAHA.109.573576. Epub 2010 Feb 18. PMID 20167912
- [Background] Brittain KR, Perry SI, Peet SM, Shaw C, Dallosso H, Assassa RP, Williams K, Jagger C, Potter JF, Castleden CM. Prevalence and impact of urinary symptoms among community-dwelling stroke survivors. Stroke. 2000 Apr;31(4):886-91. doi: 10.1161/01.str.31.4.886. PMID 10753993
- [Background] Garrett VE, Scott JA, Costich J, Aubrey DL, Gross J. Bladder emptying assessment in stroke patients. Arch Phys Med Rehabil. 1989 Jan;70(1):41-3. PMID 2916918
- [Background] Mizrahi EH, Waitzman A, Arad M, Blumstein T, Adunksy A. Bladder management and the functional outcome of elderly ischemic stroke patients. Arch Gerontol Geriatr. 2011 Sep-Oct;53(2):e125-8. doi: 10.1016/j.archger.2010.07.007. Epub 2010 Aug 12. PMID 20708280
- [Background] Mustonen S, Ala-Houhala IO, Tammela TL. Long-term renal dysfunction in patients with acute urinary retention. Scand J Urol Nephrol. 2001 Feb;35(1):44-8. doi: 10.1080/00365590151030804. PMID 11291687
- [Background] Curtis LA, Dolan TS, Cespedes RD. Acute urinary retention and urinary incontinence. Emerg Med Clin North Am. 2001 Aug;19(3):591-619. doi: 10.1016/s0733-8627(05)70205-4. PMID 11554277
- [Background] Smith MD, Seth JH, Fowler CJ, Miller RF, Panicker JN. Urinary retention for the neurologist. Pract Neurol. 2013 Oct;13(5):288-91. doi: 10.1136/practneurol-2012-000478. Epub 2013 Mar 29. PMID 23542501
- [Background] Datta SN, Chaliha C, Singh A, Gonzales G, Mishra VC, Kavia RB, Kitchen N, Fowler CJ, Elneil S. Sacral neurostimulation for urinary retention: 10-year experience from one UK centre. BJU Int. 2008 Jan;101(2):192-6. doi: 10.1111/j.1464-410X.2007.07282.x. Epub 2007 Oct 26. PMID 17970787
- [Background] Kessler TM, La Framboise D, Trelle S, Fowler CJ, Kiss G, Pannek J, Schurch B, Sievert KD, Engeler DS. Sacral neuromodulation for neurogenic lower urinary tract dysfunction: systematic review and meta-analysis. Eur Urol. 2010 Dec;58(6):865-74. doi: 10.1016/j.eururo.2010.09.024. Epub 2010 Oct 1. PMID 20934242
- [Background] Herr-Wilbert IS, Imhof L, Hund-Georgiadis M, Wilbert DM. Assessment-guided therapy of urinary incontinence after stroke. Rehabil Nurs. 2010 Nov-Dec;35(6):248-53. doi: 10.1002/j.2048-7940.2010.tb00055.x. PMID 21140719
- [Background] Tong Y, Jia Q, Sun Y, Hou Z, Wang Y. Acupuncture in the treatment of diabetic bladder dysfunction. J Altern Complement Med. 2009 Aug;15(8):905-9. doi: 10.1089/acm.2009.0062. PMID 19678782
- [Background] Yu KW, Lin CL, Hung CC, Chou EC, Hsieh YL, Li TM, Chou LW. Effects of electroacupuncture on recent stroke inpatients with incomplete bladder emptying: a preliminary study. Clin Interv Aging. 2012;7:469-74. doi: 10.2147/CIA.S37531. Epub 2012 Nov 8. PMID 23152677
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Rowe TA, Juthani-Mehta M. Diagnosis and management of urinary tract infection in older adults. Infect Dis Clin North Am. 2014 Mar;28(1):75-89. doi: 10.1016/j.idc.2013.10.004. Epub 2013 Dec 8. PMID 24484576
- [Background] Grigoryan L, Trautner BW, Gupta K. Diagnosis and management of urinary tract infections in the outpatient setting: a review. JAMA. 2014 Oct 22-29;312(16):1677-84. doi: 10.1001/jama.2014.12842. PMID 25335150
- [Background] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033
- [Background] Sagnier PP, MacFarlane G, Richard F, Botto H, Teillac P, Boyle P. Results of an epidemiological survey using a modified American Urological Association symptom index for benign prostatic hyperplasia in France. J Urol. 1994 May;151(5):1266-70. doi: 10.1016/s0022-5347(17)35229-1. PMID 7512657
- [Derived] Shin S, Lee J, Yoo J, Lim SM, Lee E. Electroacupuncture versus sham electroacupuncture for urinary retention in poststroke patients: study protocol for a multicenter, randomized controlled trial. Trials. 2016 Apr 12;17:197. doi: 10.1186/s13063-016-1315-3. PMID 27072880
- See also: The Linguistic Validation and Reliability of the Korean Version 'Qualiveen Questionnaire'. Annals of Rehabilitation Medicine. 2010 Oct;34(5):524-43. (in Korean) — http://www.komci.org/GSResult.php?RID=0041JKARM%2F2010.34.5.524&DT=6